CLINICAL TRIAL: NCT04403919
Title: Knotless Suture in Revision Total Joint Arthroplasty: A Prospective Randomized Controlled Trial
Brief Title: Knotless Suture in Revision Total Joint Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-00280
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Arthroplasty

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled trial, parallel four-arm design, single-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Revision total knee arthroplasty: control (Active Comparator)
  Interventions: Device: Conventional Closure: Knee
- Revision total knee arthroplasty: active (Experimental)
  Interventions: Device: Barbed suture closure: Knee
- Revision Total Hip Arthroplasty: control (Active Comparator)
  Interventions: Device: Conventional Closure: Hip
- Revision Total Hip Arthroplasty: active (Experimental)
  Interventions: Device: Barbed suture closure: Hip

INTERVENTIONS:
Device: Conventional Closure: Knee — Traditional closure will consist of arthrotomy (deep layer) closed with figure of eight number 1 vicryl plus followed by closure of the intermediate layer with 0 Vicryl plus. The intermediate layer will be performed at surgeon's discretion especially in thin patients. Subdermal layer with 2-0 vicryl suture followed by subcuticular 3-0 monofilament suture (monocryl PLUS, Ethicon; Johnson & Johnson) and Dermabond advanced.
  Arms: Revision total knee arthroplasty: control
Device: Barbed suture closure: Knee — The barbed suture closure will consist of number 2 Stratafix symmetric PDS PLUS for the arthrotomy, intermediate layer will be performed at surgeon's discretion in thin patients, if performed will entail stratafix spiral, subdermal 2-0 stratafix spiral monocryl plus. Followed by subcuticular 3-0 stratafix spiral monocryl plus suture and Dermabond advance.
  Arms: Revision total knee arthroplasty: active
Device: Conventional Closure: Hip — 1. The capsule will be closed with Vicryl Plus number 1
  2. Deep fascia with figure of eight interrupted number 1 braided absorbable suture (Vicryl plus, Ethicon; Johnson &Johnson, Somerville, NJ)
  3. Subdermal fat layer simple interrupted knots using number 2-0 braided absorbable sutures (Vicryl plus)
  4. Subcuticular 3-0 monofilament suture (monocryl plus , Ethicon; Johnson & Johnson)
  5. followed by the use of skin adhesive (Dermabond Advanced, Ethicon; Johnson &Johnson).
  Arms: Revision Total Hip Arthroplasty: control
Device: Barbed suture closure: Hip — 1. The capsule will be closed with stratafix symmetric PDS Plus
  2. Deep fascia will be closed with Stratafix Symmetric PDS Plus (Stratafix symmetric PDS plus, Ethicon; Johnson &Johnson, Somerville, NJ)
  3. Subdermal layer with running number 2-0 barbed suture (stratafix spiral monocryl plus, Ethicon; Johnson & Johnson, Somerville, NJ)
  4. Subcuticular suture with stratafix spiral monocryl plus, Ethicon
  5. followed by the use of skin adhesive (Dermabond advanced, Ethicon; Johnson &Johnson).
  Arms: Revision Total Hip Arthroplasty: active

SUMMARY:
Barbed suture has been demonstrated to be safe in primary hip and knee surgery and retrospective data suggests barbed suture represents no increased complications in the revision setting. Barbed suture may represent a faster, more effective way to perform revision arthroplasty closures. There are no Level I studies comparing traditional and barbed suture closure. The purpose of this study is to assess the surgical complexities of closures using closure time without sacrificing cosmesis or wound complications between the traditional closure and barbed closure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. Surgical candidates undergoing revision total knee or total hip arthroplasty for one of the following indications second stage of two stage reimplantation for infection, mechanical loosening, instability, polyethylene wear, stiffness, or periprosthetic fracture

Exclusion Criteria:

1. Patient is ≤ 18 years of age
2. Patient is unable to provide written consent
3. Patient has active infections in the operative leg/joint
4. Known Allergy to Suture material
5. Underlying Dermatological diseases affecting surgical site including dermatitis, eczema, or psoriasis; connective tissue or vascular disorders or diseases that would adversely affect wound healing; metastatic cancer; renal insufficiency (dialysis); steroid dependence; malnourishment; and other disease processes resulting in an immunocompromised state. Diabetes, smoking and obesity will be allowed as they are frequent comorbidities in our revision joint population
6. Anterior total hip replacement
7. Stage 1 of two stage revision for infection
8. Closure performed by plastic surgeon, including flap coverage

Vulnerable populations will not be enrolled in this study.

Withdrawal Criteria

1. Failure to attend regularly scheduled follow up appointments
2. Deviation from closure protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ran Schwarzkopf, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [contact information for PI or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to ran.schwarzkopf@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Revision Total Knee Arthroplasty: Control | Revision Total Knee Arthroplasty: Active | Revision Total Hip Arthroplasty: Control | Revision Total Hip Arthroplasty: Active
Started | 22 | 30 | 18 | 11
Completed | 22 | 30 | 18 | 10
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Revision Total Knee Arthroplasty: Control | Revision Total Knee Arthroplasty: Active | Revision Total Hip Arthroplasty: Control | Revision Total Hip Arthroplasty: Active | Total
Number analyzed (Participants) | 22 | 30 | 18 | 10 | 80
Age, Continuous [Mean (Full Range); unit: years] | 64.3 [53 to 80] | 63.3 [48 to 84] | 61.7 [33 to 78] | 64.9 [42 to 89] | 63.4 [33 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 14 | 5 | 53
  Male | 6 | 12 | 4 | 5 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 9 | 4 | 0 | 18
  White | 13 | 10 | 10 | 8 | 41
  More than one race | 4 | 11 | 3 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 30 | 18 | 10 | 80

OUTCOME MEASURES:

1. Primary Outcome: Time of Closure in Minutes
Description: Measurement of the time needed to properly close the wound with each technique.
Time Frame: Up to a maximum of 66 minutes (perioperative)
Measure: Mean (Full Range); unit: minutes
Groups:
- Revision Total KNEE Arthroplasty: Control (Conventional Closure): Conventional Closure: Knee: Traditional closure will consist of arthrotomy (deep layer) closed with figure of eight number 1 vicryl plus followed by closure of the intermediate layer with 0 Vicryl plus. The intermediate layer will be performed at surgeon's discretion especially in thin patients. Subdermal layer with 2-0 vicryl suture followed by subcuticular 3-0 monofilament suture (monocryl PLUS, Ethicon; Johnson & Johnson) and Dermabond advanced.
- Revision Total KNEE Arthroplasty: Active (Barbed Suture Closure): Barbed suture closure: Knee: The barbed suture closure will consist of number 2 Stratafix symmetric PDS PLUS for the arthrotomy, intermediate layer will be performed at surgeon's discretion in thin patients, if performed will entail stratafix spiral, subdermal 2-0 stratafix spiral monocryl plus. Followed by subcuticular 3-0 stratafix spiral monocryl plus suture and Dermabond advance.
- Revision Total HIP Arthroplasty: Control (Conventional Closure): Conventional Closure: Hip: 1. The capsule will be closed with Vicryl Plus number 1 2. Deep fascia with figure of eight interrupted number 1 braided absorbable suture (Vicryl plus, Ethicon; Johnson &Johnson, Somerville, NJ) 3. Subdermal fat layer simple interrupted knots using number 2-0 braided absorbable sutures (Vicryl plus) 4. Subcuticular 3-0 monofilament suture (monocryl plus , Ethicon; Johnson & Johnson) 5. followed by the use of skin adhesive (Dermabond Advanced, Ethicon; Johnson &Johnson).
- Revision Total HIP Arthroplasty: Active (Barbed Suture Closure): Barbed suture closure: Hip: 1. The capsule will be closed with stratafix symmetric PDS Plus 2. Deep fascia will be closed with Stratafix Symmetric PDS Plus (Stratafix symmetric PDS plus, Ethicon; Johnson &Johnson, Somerville, NJ) 3. Subdermal layer with running number 2-0 barbed suture (stratafix spiral monocryl plus, Ethicon; Johnson & Johnson, Somerville, NJ) 4. Subcuticular suture with stratafix spiral monocryl plus, Ethicon 5. followed by the use of skin adhesive (Dermabond advanced, Ethicon; Johnson &Johnson).
Arm/Group | Revision Total KNEE Arthroplasty: Control (Conventional Closure) | Revision Total KNEE Arthroplasty: Active (Barbed Suture Closure) | Revision Total HIP Arthroplasty: Control (Conventional Closure) | Revision Total HIP Arthroplasty: Active (Barbed Suture Closure)
Number analyzed (Participants) | 22 | 30 | 18 | 10
minutes | 36.3 [18.7 to 51.0] | 31.1 [17.3 to 45.0] | 35.9 [17.5 to 66.0] | 27.1 [18.7 to 47.0]

2. Secondary Outcome: Incidence of Complications Related to Wound Closure
Description: Number of all complications (including needle sticks and glove perforations) and infections related to the wound closure.
Time Frame: Day 90
Measure: Number; unit: Total number of complications
Arm/Group | Revision Total KNEE Arthroplasty: Control (Conventional Closure) | Revision Total KNEE Arthroplasty: Active (Barbed Suture Closure) | Revision Total HIP Arthroplasty: Control (Conventional Closure) | Revision Total HIP Arthroplasty: Active (Barbed Suture Closure)
Number analyzed (Participants) | 22 | 30 | 18 | 10
Total number of complications | 2 | 4 | 1 | 0

3. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS) Score
Description: The POSAS consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically on a ten-step scale, where 0 = normal skin and 10 = worst scar imaginable. Together they make up the 'Total Score' of the Patient and Observer Scale, which ranges from 0 to 120; higher scores indicate worse scars.
Time Frame: Week 6 Post-Surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Revision Total KNEE Arthroplasty: Control (Conventional Closure) | Revision Total KNEE Arthroplasty: Active (Barbed Suture Closure) | Revision Total HIP Arthroplasty: Control (Conventional Closure) | Revision Total HIP Arthroplasty: Active (Barbed Suture Closure)
Number analyzed (Participants) | 22 | 30 | 18 | 10
score on a scale | 2.7 [1.0 to 4.0] | 3.4 [1.0 to 5.0] | 2.5 [1.0 to 5.0] | 2.6 [1.0 to 4.0]

4. Secondary Outcome: Mean Number of Sutures Used
Time Frame: 45 minutes (perioperative)
Measure: Mean (Full Range); unit: sutures
Arm/Group | Revision Total KNEE Arthroplasty: Control (Conventional Closure) | Revision Total KNEE Arthroplasty: Active (Barbed Suture Closure) | Revision Total HIP Arthroplasty: Control (Conventional Closure) | Revision Total HIP Arthroplasty: Active (Barbed Suture Closure)
Number analyzed (Participants) | 22 | 30 | 18 | 10
sutures | 10.9 [4.0 to 15.0] | 6.3 [4.0 to 10.0] | 9.1 [5.0 to 12.0] | 5.9 [4.0 to 8.0]

5. Secondary Outcome: Mean Length of Incision
Time Frame: 30 minutes (perioperative)
Measure: Mean (Full Range); unit: millimeters
Arm/Group | Revision Total Knee Arthroplasty: Control | Revision Total Knee Arthroplasty: Active | Revision Total Hip Arthroplasty: Control | Revision Total Hip Arthroplasty: Active
Number analyzed (Participants) | 22 | 30 | 18 | 10
millimeters | 196.4 [145 to 300] | 186 [110 to 290] | 168 [120 to 230] | 177 [135 to 240]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Revision Total KNEE Arthroplasty: Control (Conventional Closure) | Revision Total KNEE Arthroplasty: Active (Barbed Suture Closure) | Revision Total HIP Arthroplasty: Control (Conventional Closure) | Revision Total HIP Arthroplasty: Active (Barbed Suture Closure)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/30 | 0/18 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/22 | 2/30 | 0/18 | 0/11
Other Adverse Events (participants affected / at risk) | 1/22 | 2/30 | 1/18 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revision Total KNEE Arthroplasty: Control (Conventional Closure) (N=22) | Revision Total KNEE Arthroplasty: Active (Barbed Suture Closure) (N=30) | Revision Total HIP Arthroplasty: Control (Conventional Closure) (N=18) | Revision Total HIP Arthroplasty: Active (Barbed Suture Closure) (N=11)
Recurrent effusion (Infections and infestations) | 1 | 0 | 0 | 0
Traumatic wound dehisence (General disorders) | 0 | 1 | 0 | 0
Lateral capsule weekness and herniation (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revision Total KNEE Arthroplasty: Control (Conventional Closure) (N=22) | Revision Total KNEE Arthroplasty: Active (Barbed Suture Closure) (N=30) | Revision Total HIP Arthroplasty: Control (Conventional Closure) (N=18) | Revision Total HIP Arthroplasty: Active (Barbed Suture Closure) (N=11)
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Delayed wound healing (General disorders) | 0 | 1 | 0 | 0
Instability/Dislocation (General disorders) | 0 | 0 | 0 | 1
Recurrent effusion (Infections and infestations) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT04403919/Prot_SAP_000.pdf